Date: April 18th, 2017

Project Title: Studies of Growth Deficiency and Growth Hormone Treatment in Children with Osteogenesis Imperfecta Types III and IV

Principal Investigator: Joan C. Marini, M.D., Ph.D. Chief, Bone and Extracellular Matrix Branch, NICHD, NIH

## **Statistical Analysis Plan:**

For each patient, they were seen at the NIH CC for a full year prior to treatment.

**Baseline growth rate** was set for each patient at NIH CC: At 1 yr prior and 6 months prior to treatment, as well as at t=0, patients length was measured on a stadiometer board by genetics and endocrine nurses trained to take accurate repetitive measurements. 10 measurements were taken and averaged for each date. The growth in cc from 1 year prior to treatment to treatment start in cm/yr was the baseline growth rate for that patient.

**Treatment growth rate:** Measurements taken on each patient at treatment time=0, 6 and 12 months were taken in the same way and a treatment year (cm/yr) growth rate was calculated.

**Response to treatment:** For each patient, their rate of growth during treatment was compared to the baseline growth rate. A positive response was scored if treatment growth rate was 50% or more increased over baseline rate. The percent of patients in the full treatment group with a positive linear growth rate response was scored as the % responders.